CLINICAL TRIAL: NCT07038304
Title: Oligometastatic Directed Radiotherapy for Patients With Castration Resistant Prostate Cancer
Brief Title: The Impact of Metastatic Directed Radiotherapy (MDRT) on Oligoprogressive Castration Resistant Prostate Cancer (CRPC)
Acronym: OLYMPIAN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL87430.042.24
Record Dates: First submitted 2025-03-04; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer (Adenocarcinoma); OligoProgressive Metastatic Disease; Castration Resistant Metastatic Prostate Cancer; Radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MDRT to oligoprogression (Experimental): Patients included in the study with a post prostatectomy local recurrence on the PSMA PET with up to 3 oligometastases will be treated preferably with SBRT to all oligometastatic lesions and to the local recurrence in prostate bed
  Interventions: Radiation: Metastasis directed radiotherapy

INTERVENTIONS:
Radiation: Metastasis directed radiotherapy — According to guidelines, in the case of oligoprogression next line systemic treatment is recommended. This study investigates the potential delay of NEST and rPFS by MDRT.

SUMMARY:
In patients with metastatic prostate cancer (PCa) who receive androgen deprivation therapy (ADT), the sensitivity to castration will eventually disappear due to the selection of castration-refractory clones. This will lead to the stage of metastatic castration-refractory prostate can-cer (mCRPC), which is incurable and results in a median overall survival of 2-3 years.

Treatment options for patients with mCRPC include several systemic agents, such as andro-gen receptor-targeted agents (ARTA), chemotherapy (docetaxel, cabazitaxel) and bone-targeting agents (radium- 223). Clinical progression and, to a lesser extent, biochemical pro-gression traditionally imply a switch to the next line systemic treatment (NEST). Within patients with mCRPC, there is a subgroup showing oligo-progression, defined as the progression of up to 3 lesions, including both metastatic and/or local relapse. Oligoprogression reflects a heterogeneous treatment response, which, in turn, reflects the heterogeneity of the clonogenic cells that give rise to mCRPC. Retrospective studies suggest that metastasis-directed radiotherapy (MDRT) to these oligoprogressive lesions delayed the need for NEST. Recently, promising results were published on the use of MDRT in the oligopro-gressive mCRPC (omCRPC) setting, with a NEST-free survival (NEST-FS) of 21 months in well selected patients. Currently, in The Netherlands, patients with omCRPC are frequently referred and treated with MDRT, but a clear treatment protocol and inclusion/selection criteria are missing. Moreover, the exact benefit of MDRT in patients with omCRPC remains unclear, as prospective evi-dence for MDRT in omCRPC is lacking.

DETAILED DESCRIPTION:
The primary aim of this study is to test the hypothesis that the addition of MDRT to standard of care (ADT or ADT + chemotherapy or ARTA) in well-selected PCa patients with oligometastatic progressive disease, defined on PSMA PET, prolongs the radiological progression-free survival (rPFS) and postpones the start of next line systemic therapy (NEST). Patients included in this study already have an indication to start NEST, and any delay introduced by adding MDRT will result in a net benefit for the patients.

Primary objectives include: Postponement of the start of next line systemic treatment (NEST), and enhancement of the radiological progression-free survival (rPFS) In this single arm multicenter prospective phase II trial, we aim to include 35 patients with omCRPC (1-3 metastases and/or local recurrence) who will be treated with MDRT to the visible progressive lesions (up to max of 3). Progression is based on PSMA PET.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the prostate.
* mCRPC setting, with testosterone level < 50 ng/dl or 1.7 nmol/l.
* Oligoprogressive disease diagnosed on PSMAscan; defined as the progression of pre-existing metastatic disease, and/or the appearance of new metastases and/or the appearance of a local relapse with a maximum of 3 lesions in total.
* Patients currently treated with ADT, whether combined with another systemic treatment such as ARTA, chemotherapy.
* For patients treated with chemotherapy, the course should be completed or stopped before start MORT - In case of treatment with ARTA, a minimal of 3 months response (PSA or clinical response).
* WHO performance status 0-2.
* Age > = 18 years old.
* Patiënt should be presented at the multidisciplinary tumor board of the local hospital in which the therapy will be given.
* Before patiënt registration, written informed consent must be given according to ICH/GCO and national/local regulations.

Exclusion Criteria:

* Serum testosterone level > 50 ng/ml or > 1.7 nmol/l.
* Presence of more than 3 progressive/new metastatic lesions and/or local recurrence (which counts for 1 lesion).
* Active malignancy other than prostate cancer that can potentially interfere with the interpretation of the trial, except non-melanoma skin cancer or non-invasive urothelial cell carcinoma.
* Local recurrence in the prostate after previous radiotherapy
* Previous treatments (RT, surgery) or comorbidities making new treatment with MDRT impossible.
* Disorder precluding understanding of trial Information or informed consent or signing informed consent.
* Evidence of PSMA-negative disease.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer is limited to males.
Enrollment: 35 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2028-01-03 (Estimated); Study Completion 2029-01-03 (Estimated)

PRIMARY OUTCOMES:
NEST-FS | 6, 12-and 24-months
  Next line systemic treatment free survival
rPFS | 6, 12-and 24-months
  radiologic progression free survival

SECONDARY OUTCOMES:
Quality of Life (QoL) | baseline, 6 months, 12 months, 24 months
  Evaluated using the EORTC QLQ-C30 for health related QoL.
Biochemical progression | From date of randomization until the date of first documented biochmical progression, assessed up to 36 months
  after an initial decline in PSA: the time from start of therapy to first PSA increase that is ≥25% and ≥ 2 ng/ml above the nadir, and which is confirmed by a second value ≥3 weeks later.
Overall survival (OS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  Overall survival
Quality of life (QoL) | baseline, 6 months, 12 months, 24 months
  EORTC PR-25 for prostate symptom specific QoL.
Acute grade ≥ 2 gastrointestinal toxicity | Up to 3 months after completion of the RT
  As assessed using physician-reported score: Common Terminology Criteria for adverse events version 5.0 (CTCAE-5) toxicity score with a scale of 1 - 4.
Acute grade ≥ 2 gastrointestinal toxicity | Up to 3 months after completion of the RT
  Using patient-reported questionnaires (Radiation Therapy Oncology Group (RTOG) / European platform of cancer research (EORTC) toxicity questionnaires with grade 1 to 4).
Acute grade ≥ 2 genitourinary toxicities | Up to 3 months after completion of the RT
  As assessed using physician-reported score using questionnaires (CTCAE 5.0 toxicity score).
Acute grade ≥ 2 genitourinary toxicities | Up to 3 months after completion of the RT
  Using patient-reported questionnaires (Radiation Therapy Oncology Group (RTOG) / European platform of cancer research (EORTC) toxicity questionnaires with grade 1 to 4).
Late grade ≥ 2 genitourinary toxicities | Up to 2 years after completion of the RT
  Using patient-reported questionnaires (Radiation Therapy Oncology Group (RTOG) / European platform of cancer research (EORTC) toxicity questionnaires with grade 1 to 4).
Late grade ≥ 2 genitourinary toxicity | Up to 2 years after completion of the RT
  Using physician-reported score (CTCAE 5.0 toxicity score).
Late grade ≥ 2 gastrointestinal toxicity | Up to 2 years after completion of the RT
  As assessed using physician-reported score (CTCAE 5.0 toxicity score).
Late grade ≥ 2 gastrointestinal toxicity | Up to 2 years after completion of the RT
  Using patient-reported questionnaires (Radiation Therapy Oncology Group (RTOG) / European platform of cancer research (EORTC) toxicity questionnaires with grade 1 to 4).

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - UMC Groningen, Groningen
  - Radboud Umc, Nijmegen